CLINICAL TRIAL: NCT06356454
Title: Knowledge, Attitudes and Practices of Paediatric Cardiologists About Cardiac Rehabilitation in Children With Congenital Heart Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Haluk Tekerlek, Research assistant, PhD, Karamanoğlu Mehmetbey University
Other Study IDs: KAPCON-CR
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Physician's Role

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire on knowledge, attitudes and practices of paediatric cardiologists about cardiac rehabilitation in children with congenital heart disease — Creating the questionnaire: The self-administered questionnaire was designed based on literature review. The questions of the questionnaire were based on the 3 main components of the World Health Organisation's Knowledge, Attitude and Practice framework. The questions were evaluated by experts in the field such as cardiologists working in paediatric cardiology. The questionnaire, which was finalised with the questions updated according to expert opinions, has 5 sections:
  * Section 1: Socio-demographic questions
  * Section 2: Questions on the level of knowledge about CR
  * Section 3: Questions on attitudes about CR
  * Section 4: Questions on Practices about CR

SUMMARY:
Despite significant clinical benefits and recommendations of clinical practice guidelines to refer patients for exercise and physical activity counselling in the capacity of cardiac rehabilitation (CR), CR is largely underutilised and not implemented effectively. Studies have reported that the reasons for the low implementation of CR are multifactorial at the healthcare system, physician and patient levels. Therefore, the aim of this study was to investigate the knowledge, attitudes and practical applications of paediatric cardiologists regarding cardiac rehabilitation and specifically exercise and physical activity in children with congenital heart disease (CHD).

ELIGIBILITY:
Inclusion Criteria:

* To be a paediatric cardiologist,
* Providing active service in patient diagnosis and treatment

Exclusion Criteria:

* Not providing active service in patient diagnosis and treatment despite being a paediatric cardiologist (administrative position, etc.).

Ages: 32 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study is paediatric cardiologists. The sample consists of paediatric cardiologists who volunteered to participate in the study, to whom the study could be announced/notified, and who actively serve in patient diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-02 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
The score of Questionnaire on knowledge, attitudes and practices of paediatric cardiologists about cardiac rehabilitation in children with congenital heart disease | 10-15 minutes
  The scale created in this study does not have a minimum and maximum score due to its nature. Some questions in the scale are in yes/no format and some questions are in multiple choice format. For this reason, the results of the study will be given in the form of categorical or frequency tables in accordance with the scale questions. The questions consist of knowledge of physicians about CR, attitudes of physicians on CR, practices of physicians on CR and barriers faced by physicians for referring to CR and socio-demographic data of the responders.

IPD SHARING:
Plan to Share IPD: Undecided